CLINICAL TRIAL: NCT04403490
Title: Effect of Hand and Arm Bimanual Intensive Therapy Including Lower Extremities on the Body Function and Structures of Children With Bilateral and Unilateral Cerebral Palsy, Including Selective Voluntary Motor Control and Brain Structure
Brief Title: Effect of HABIT-ILE on the Body Function and Structures of Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B403201316810f
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: motor skill learning; body function; body structure; selective voluntary motor control; brain structure; neuroplasticity; intensive therapy; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE (Experimental): Hand and arm bimanual intensive therapy including lower extremities
  Interventions: Behavioral: HABIT-ILE
- Conventional intervention (Active Comparator): Conventional physical and occupational therapy
  Interventions: Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: HABIT-ILE — 2 weeks HABIT-ILE
  Arms: HABIT-ILE
Behavioral: Conventional intervention — 2 weeks usual intervention (waitlist group)
  Arms: Conventional intervention

SUMMARY:
There is strong evidence that recent intensive interventions based on motor skill learning principles are efficient on functional and neuroplastic changes of children with cerebral palsy (CP).

Besides, impaired selective voluntary motor control (SVMC) is one of four interrelated neuromuscular deficits in children with CP and is listed in the ICF-CY (International Classification of Functioning, Disability and Health for Children and Youth) under body functions. Additionally, impaired SVMC has been shown to negatively affect the motor and functional abilities of children with CP. However, there have been little scientific investigations on the trainability of SVMC according to therapeutic interventions.

Therefore, the study aims to evaluate the effect of Hand and Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) on the body function and structures of children with bilateral and unilateral cerebral palsy, including SVMC and brain structure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed bilateral and unilateral cerebral palsy,
* MACS levels from I to IV,
* GMFCS levels from I to IV,
* Ability to follow instructions and complete testing.

Exclusion Criteria:

* Orthopedic surgery, botulinum toxin injections or another unusual intervention less than 6 months before or within the study period.
* Unstable seizure
* Severe visual or cognitive impairments likely to interfere with intervention or testing session completion

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Diffusion Tensor Imaging (DTI) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  This sequence allows to measure changes in the fractional anisotropy (FA) on the white matter tracts. FA is a scalar value (no unit) between zero and one that describes the degree of anisotropy of white matter water molecules.
Changes in Test of Arm Selective Control (TASC) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The TASC is an upper limb selective motor control evaluation tool including eight motions in each arm and up to three attempts are allowed for each motion. This assessment tool was developed in 2010 and Sukal-Moulton et al. have proved its validity and reliability for children with CP in 2017. After completion of the best attempt, points ranging from 0 (absent), 1 (impaired) to 2 (normal) are recorded for each joint depending on the movement properties and descriptors of the test.
Changes in Selective Control Assessment of the Lower Extremity (SCALE): | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The SCALE was designed to evaluate lower limb selective motor control of children with cerebral palsy. The SCALE includes testing of five reciprocal lower extremity movements. SVMC is graded at each joint as 'Normal' (2 points), 'Impaired' (1 point), or 'Unable' (0 points).
Changes in Strength | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The strength will be measured for main muscle groups using a Microfet.
Changes in Stiffness | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The stiffness will be measured using a device developed and already validated at UCLouvain.

SECONDARY OUTCOMES:
Changes in Assisting Hand Assessment (AHA or BoHA) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The AHA is a videotaped tool measuring how effectively children with unilateral CP use the affected hand in bimanual activities. The BoHA is a videotaped tool measuring how effectively children with bilateral CP use both hands in bimanual activities.
Changes in ABILHAND-Kids Questionnaire | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The ABILHAND-Kids Questionnaire has been developed to assess a child's unimanual and bimanual upper limb activities. It ranges from - 6 to +6 logits (higher score means better performance).
Changes in ACTIVLIM-CP Questionnaire | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The ACTIVLIM-CP Questionnaire measures a patient's ability to perform daily activities requiring the use of the upper and/or the lower limbs through 42 items specific to patients with cerebral palsy. It ranges from - 5 to +5 logits (higher score means better performance).
Changes in Gross Motor Function Measurement (GMFM 66) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The GMFM has been developed to measure the change in gross motor function over time in children with cerebral palsy.
Changes in 6 Minutes Walking Test (6MWT) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The 6 Minutes Walking Test measures the distance that the patient walk as much as possible within a period of 6-minutes in a 30 meters long corridor.
Changes in Box and Blocks test | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The BBT is a test of gross manual dexterity. Each hand is tested individually and the BBT is scored through the number of blocks carried over the partition from one part to another part of a box during the one-minute trial period.
Changes in Jebsen-Taylor Test | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The Jebsen-Taylor Test assesses uni-manual hand function, through 7 subtests simulating daily life activities. The test assesses speed, not quality of performance and time to complete each activity is reported using a stopwatch.
Changes in Modified Cooper test | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The Modified Cooper test is a modified version of The Manual Form Perception Test, which evaluates stereognosis through 16 objects. Both hands are tested separately and time to recognise the objects is reported using a stopwatch.
Changes in ABILOCO-Kids Questionnaire | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The ABILOCO-Kids Questionnaire measures a patient's ability to perform daily activities requiring the use of the lower limbs through 10 items specific to patients with cerebral palsy. It ranges from - 4 to +4 logits (higher score means better performance).
Changes in Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The PEDI-CAT is the new version of the Pediatric Evaluation of Disability Inventory (PEDI). The PEDI-CAT is comprised of 276 functional activities acquired throughout infancy, childhood and young adulthood. Based on the nternational Classification of Functioning, Disability and Health for Children and Youth (ICF-CY) model, the PEDI-CAT contents provide information about the activities and participation component. It ranges from 0 to 100% (higher score means better performance).
Changes in Canadian Occupational Performance Measure (COPM) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The COPM measures the patient's self-perception of occupational performance and satisfaction of it in daily activities over time. It ranges from 1 to 10, a higher score means a better performance.
Changes in Double Inversion Recovery (DIR) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  This sequence allows to identify an inflamatory lesion.
Changes in Functional resting state (RS) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  This sequence allows to evaluate the regional interactions that occur in a resting or task-negative state.
Changes in T1-weighted and T2-weighted structural imaging | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The difference between these sequences allows to evaluated changes in the cortical myelin.
Changes in Executive Functions | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Cognitive functions of the children will be assessed by Stroop task and Flanker task.
Changes in spatial parameters of the gait (Kinematics assessments) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the stride length (meters), step length (meters) and step width (meters).
Changes in temporal parameters of the gait (Cycle time) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the cycle of gait time (seconds).
Changes in temporal parameters of the gait (Stance time) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the stance time (percentage of the total gait cycle).
Changes in temporal parameters of the gait (Swing time) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the swing time (percentage of the total gait cycle).
Changes in temporal parameters of the gait (Stride) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the gait cadence (stride per minute).
Changes in temporal parameters of the gait (Velocity) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the gait velocity (meter/second).
Changes in temporal parameters of the gait (Acceleration) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the gait acceleration (meters/second^2)
Changes in spatial parameters of the upper extremity (Straightness) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the straightness (percentage of upper extremity trajectory during a reaching task).
Changes in spatial parameters of the upper extremity (Smoothness) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the smoothness (variability of the movement during a reaching task)
Changes in temporal parameters of the upper extremity (Kinematics assessments) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the time from onset to end of the task (seconds). the task consists in a bimanual reaching task.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, Principal Investigator — Institute of Neuroscience, UCLouvain
Locations (1):
- Institute of Neuroscience, UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No